CLINICAL TRIAL: NCT04303624
Title: Exploring Family vs. Individual Decision-making in Organ Donation
Brief Title: Understanding Family Refusal
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Other Study IDs: HSS-1502-P02-06
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Brain Death; Renal Failure
Keywords: Organ donation; Transplantation; Intensive care
MeSH Terms: conditions — Brain Death; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community sample: Representative sample of the Singapore population
  Interventions: Other: Health sciences survey

INTERVENTIONS:
Other: Health sciences survey — Large scale demographic survey evaluating attitudes of population towards organ donation for the self vs. family

SUMMARY:
The investigators plan a secondary data analysis of an existing dataset to examine how individual decision-making differs from family decision-making in organ donation.

ELIGIBILITY:
Inclusion Criteria:

* Citizens or permanent residents of Singapore
* Above 21

Exclusion Criteria:

- Below 21

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were a representative sample of Singapore's population, approached via door-to-door recruitment and via community eateries.
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Willingness to donate | Single measurement (time of taking the survey)
  Participants indicated their willingness to donate their own organs and those of a close family member

SECONDARY OUTCOMES:
Confidence in family decision-making | Single measurement (time of taking the survey)
  Participants rated how confident they were that - upon their family member's death - they would respect their family member's views regarding donation rated using 5-point scales anchored on one end with 1="Not confident at all" and 5="Absolutely confident").

IPD SHARING:
Plan to Share IPD: No
Due to stipulations by the Institutional Review Board, there is no data that can be shared.